CLINICAL TRIAL: NCT01125540
Title: The Role of Daily Disposable Contact Lenses in Ocular Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: National Pollen and Aerobiology Unit, Worcester (Unknown)
Responsible Party: Prof James Wolffsohn, Aston University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Allergy02
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Grass Pollen Ocular Allergy
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Acuvue (Standard Daily Disposable Contact Lens)
  Other Names: Acuvue
Device: CIBA Dailies Aquacomfort Plus (Contact Lens - enhance lubricating)
  Other Names: CIBA Dailies Aquacomfort Plus

SUMMARY:
Patients with seasonal allergic conjunctivitis are normally advised to avoid contact lens wear when they are having symptoms. However, modern soft contact lenses which are disposed of daily offer the potential to protect and lubricate the ocular surface. This study examines this possible effect.

ELIGIBILITY:
Inclusion Criteria:

* contact lens wearer
* proven allergy to grass pollen

Exclusion Criteria:

* eye disease
* ocular medication
* allergy medication
* asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Symptoms | 4 hours
  Subjective rating of itchyness, dryness, burning, watering and discomfort
Signs | 4 hours
  Signs of bulbar, limbal and palpebtal hyperaemia and staining

CONTACTS AND LOCATIONS:
Locations (1):
- Aston University, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Wolffsohn JS, Emberlin JC. Role of contact lenses in relieving ocular allergy. Cont Lens Anterior Eye. 2011 Aug;34(4):169-72. doi: 10.1016/j.clae.2011.03.004. Epub 2011 May 6. PMID 21530362